CLINICAL TRIAL: NCT06468280
Title: Synergistic Effects of PD-1 Antibody and Chemotherapy/Targeted Therapy Followed by Surgery-centric Local Treatment in Patients With Limited-metastatic Gastric or Gastroesophageal Adenocarcinoma (ROSETTE Trial): an Open-label, Single-center, Randomized Phase 2 Trial
Brief Title: Synergistic Effects of PD-1 Antibody and Chemotherapy/Targeted Therapy Followed by Surgery-centric Local Treatment in Patients With Limited-metastatic Gastric Cancer
Acronym: ROSETTE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xuefei.Wang, Chief of Gastrointestinal Surgery Department, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2024164
Record Dates: First submitted 2024-05-28; First posted 2024-06-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer; GastroEsophageal Cancer
Keywords: Limited metastasis; Surgery; Local treatment; Gastric cancer; Perioperative treatment
MeSH Terms: conditions — Stomach Neoplasms | interventions — Surgical Procedures, Operative; spartalizumab; Trastuzumab; zolbetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local Treatment Arm (Arm A) (Experimental): In Phase 1, patients will receive four cycles of PD-1 antibody in combination with chemotherapy, with or without targeted therapy. Following this phase, a radiologic assessment will evaluate disease progression status. Patients identified as not experiencing progression will proceed with the study treatments. Subsequently, they will undergo surgeon-led local treatment, which may include standard D2 gastrectomy and metastasectomy when feasible. Non-surgical local treatments may also be administered to address unresected or unresectable metastatic lesions, either concurrently or sequentially with surgery. After surgical intervention, patients will receive up to four additional cycles of treatment, followed by maintenance therapy during Phase 2 of the systemic treatment. The total treatment duration may extend up to two years from the date of enrollment.
  Interventions: Procedure: Local treatment (Surgical); Drug: PD-1 Monoclonal Antibody; Drug: XELOX/SOX Chemotherapy Regimen; Procedure: Local Treatment (Non-surgical); Drug: Trastuzumab; Drug: Zolbetuximab
- Systemic Treatment Arm (Arm B) (Active Comparator): In Phase 1, patients will receive four cycles of PD-1 antibody in conjunction with chemotherapy, with or without targeted therapy. Following this phase, a radiologic assessment will evaluate the disease progression status. Patients classified as not experiencing progression-defined as the absence of local progression, advancement of existing distant metastases, or the emergence of new distant metastatic lesions-will continue with the study treatments. In Phase 2, participants will receive an additional up to four cycles of treatment, followed by maintenance therapy. The total treatment duration could extend up to two years from the date of enrollment.
  Interventions: Drug: PD-1 Monoclonal Antibody; Drug: XELOX/SOX Chemotherapy Regimen; Drug: Trastuzumab; Drug: Zolbetuximab

INTERVENTIONS:
Procedure: Local treatment (Surgical) — Radical gastrectomy with standard D2 lymphadenectomy will be performed, along with radical surgery for resectable metastatic lesions.
  Arms: Local Treatment Arm (Arm A)
Drug: PD-1 Monoclonal Antibody — PD-1 monoclonal antibody will be administered at a dosage of 200 mg via intravenous infusion (or according to the prescribing information of specific drug), once every cycle, each cycle spanning three weeks. The specific PD-1 antibody used will be determined by the investigators based on clinical considerations. Potential options include Sintilimab, Tislelizumab, or other approved PD-1 antibody products indicated for the treatment of metastatic gastric or gastroesophageal adenocarcinoma.
Drug: XELOX/SOX Chemotherapy Regimen — Oxaliplatin: 130 mg/m² administered via a 3-hour intravenous infusion on D1 of each 3-week cycle.
  Capecitabine: 1000 mg/m² taken orally twice daily. The first dose is administered on the evening of D1, and the last dose on the morning of D15, consisting of 2 weeks of treatment and a 1-week break in each 3-week cycle.
  S-1: 40 mg/m² taken orally twice daily. The first dose is administered on the evening of D1, and the last dose on the morning of D15, consisting of 2 weeks of treatment and a 1-week break in each 3-week cycle.
  During the maintainance phase, only capecitabine/S-1 will be administered.
Procedure: Local Treatment (Non-surgical) — Additional local treatment for unresected metastatic lesions during phase 2 systemic therapy is permitted, including:
  * Bone metastasis, distant lymph nodes, adrenal metastasis: Radiation therapy.
  * Lung and liver metastasis: Radiofrequency ablation, interventional embolization, or radiation therapy.
  * Peritoneal metastasis: Hyperthermic intraperitoneal chemotherapy (HIPEC).
  * Other metastatic lesions: Non-surgical treatment options discussed by the multidisciplinary team.
  Arms: Local Treatment Arm (Arm A)
Drug: Trastuzumab — For HER2-positive patients, the dosing regimen for the addition of trastuzumab is as follows:
  During the combination phase with XELOX/SOX chemotherapy: 8 mg/kg administered as an intravenous infusion on D1.
  During the maintenance phase with capecitabine/S-1: 6 mg/kg administered as an intravenous infusion on D1.
  This is repeated once every 3 weeks.
Drug: Zolbetuximab — For patients with Claudin18.2-positive expression (IHC 2-3+ in ≥75% of tumor cells), Zolbetuximab may be added with the following dosing regimen:
  First cycle: 800 mg/m² administered as an intravenous infusion on D1. Subsequent cycles: 600 mg/m² administered as an intravenous infusion on D1. This is repeated once every 3 weeks.

SUMMARY:
ROSETTE trial is an open-label, randomized phase II study designed to investigate treatment strategies for patients with limited metastatic gastric or gastroesophageal adenocarcinoma. Eligible patients are randomized to receive either systemic treatment followed by surgeon-led local treatment, or systemic treatment alone. Systemic treatment combines immunotherapy with chemotherapy, with or without targeted therapy, while the surgeon-led local treatment utilizes a surgery-centric, multi-modality approach involving resection of both primary and metastatic tumors where feasible. For unresected or unresectable metastatic lesions, alternative local therapies are provided. The primary endpoint is the 1-year event-free survival (EFS) rate. Secondary endpoints include objective response rate (ORR), disease control rate (DCR), extended EFS, overall survival (OS), pathologic complete response rate (pCR), major pathologic response rate (MPR), and R0 resection rate.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18-79.
2. Pathologically confirmed gastric adenocarcinoma or gastroesophageal junction adenocarcinoma (Siewert II or III only) with known PD-L1 expression status.
3. Gastric cancer with proficient mismatch repair (pMMR) or microsatellite stability (MSS) as determined by immunohistochemistry or NCI-recommended microsatellite markers.
4. Primary gastric cancer lesions are resectable, with limited distant metastases meeting the either of the following criteria: (1) condition (a) only; (2) any single condition from (b), with or without (a).

   (a) Non-regional intra-abdominal lymph node metastasis: Include metastasis to the superior mesenteric artery, middle colic artery, and para-aortic/retroperitoneal nodes (according to AJCC 8th edition standards).

   (b1) Localized peritoneal metastasis: P0CY1, P1a, or P1b, according to the Japanese Classification of Gastric Carcinoma (15th edition).

   (b2) Liver metastasis: Up to 5 metastatic lesions. (b3) Lung metastasis: Up to 5 unilateral metastatic lesions. (b4) Ovarian metastasis: Unilateral or bilateral. (b5) Adrenal metastasis: Unilateral or bilateral. (b6) Single-region extra-abdominal lymph node metastasis: Such as cervical, supraclavicular, or mediastinal lymph nodes.

   (b7) Bone metastasis limited to a single radiation field. (b8) Other limited metastases as determined by the research team.
5. No previous anti-tumor treatments.
6. ECOG score ≤2, no surgical contraindications.
7. Life expectancy ≥ 3 months.
8. Physical condition and organ function suitable for major abdominal surgery.
9. Willingness and ability to comply with the study protocol.
10. Fertile women with a negative urine or serum pregnancy test and agreement to use effective contraception during the study and for 180 days after the last dose. Non-sterilized men must also agree to use effective contraception.
11. Signed informed consent with an understanding that patients can withdraw anytime.

Exclusion Criteria:

1. Inability to tolerate oral chemotherapy.
2. Primary gastric lesion confined to the mucosa or submucosa with isolated ovarian metastasis.
3. Central nervous system metastasis and/or carcinomatous meningitis.
4. Allergy to any components of the study medication.
5. History of previous malignancies or concurrent other malignancies, with the exception of completely resected basal cell or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast, and other tumors with no recurrence for at least 5 years.
6. Uncontrolled pleural effusion, pericardial effusion, or ascites.
7. Weight loss ≥20% within two months before enrollment.
8. Upper gastrointestinal obstruction or physiological dysfunction.
9. Previous cytotoxic chemotherapy, radiotherapy, immunotherapy, or curative surgery.
10. Prior PD-1/PD-L1/PD-L2 or other T-cell-targeting therapy.
11. Systemic steroid or immunosuppressant use within 14 days before enrollment.
12. Live vaccine within four weeks prior to enrollment.
13. Uncontrolled systemic disease.
14. Active or past autoimmune diseases that may recur.
15. Severe chronic infections or active infections requiring systemic antibacterial, antifungal, or antiviral treatment.
16. History of lung disease.
17. Pregnancy, lactation, or planning for pregnancy.
18. HBsAg-positive with HBV DNA ≥500 IU/mL.
19. Positive HIV antibody.
20. Conditions that may impact study compliance or participation.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) Rate | 1 year from the time of randomization
  Defined as the time from randomization to the first occurrence of any event, including disease progression (local progression, local recurrence, progression of existing distant metastatic lesions, or the emergence of new distant metastases) or death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From randomization to the date of completing phase 1 systemic treatment, an average of 12 weeks.
  The proportion of subjects achieving complete response (CR) or partial response (PR) after completing phase I systemic treatment.
Disease Control Rate (DCR) | From randomization to the date of completing phase 1 systemic treatment, an average of 12 weeks.
  The proportion of subjects achieving CR, PR, or stable disease (SD) after completing phase I systemic treatment.
Pathological Complete Response (pCR) Rate | From randomization to the date of surgery, an average of 14 weeks.
  The proportion of surgical cohort subjects with no residual tumor cells and no positive lymph nodes (ypT0N0) in the primary tumor specimen. Non-surgical subjects in the surgical cohort are considered non-pCR.
Major Pathologic Response Rate (MPR) | From randomization to the date of surgery, an average of 14 weeks.
  The proportion of surgical cohort subjects with residual tumor cells <10% in the primary tumor specimen based on the Becker tumor regression grading (TRG) standard (1a-1b). Non-surgical subjects in the surgical cohort are considered non-MPR.
R0 Resection Rate | From randomization to the date of surgery, an average of 14 weeks.
  R0 resection is defined as no tumor at the gross or microscopic resection margins following standard D2 lymphadenectomy gastrectomy.
Overall Survival (OS) | Up to 5 years follow-up
  Time from randomization to death from any cause. Survivors are censored at the last known survival date.
Event-Free Survival (EFS) | Up to 5 years follow-up
  Time from randomization to the first occurrence of disease progression (local recurrence, new distant metastasis, or progression of existing metastases) or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xuefei Wang, MD, PhD, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai City
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu YY, Lee LC, Zeng H, Gu Y, Xu C, Chen WD, Shen ZB, Shen KT, Cui YH, Sun YH, Liu TS, Tang ZQ, Wang XF. Synergistic effects of PD-1 antibody and chemotherapy followed by surgery-centric local treatment in patients with limited-metastatic gastric or gastroesophageal adenocarcinoma (ROSETTE trial): an open-label, single-center, randomized phase 2 trial. BMC Cancer. 2025 Jun 1;25(1):981. doi: 10.1186/s12885-025-14331-5. PMID 40452026